CLINICAL TRIAL: NCT01390649
Title: An Open-label, Prospective, Multicenter Study to Investigate the Specificity of in Vivo Antibody Binding to Red Blood Cells in Subjects With Chronic Immune Thrombocytopenic Purpura (ITP) Treated With IgPro10 (Privigen®) Who Have Shown Signs of Hemolysis
Brief Title: A Safety Study of Intravenous Immunoglobulin in Patients With Chronic Immune Thrombocytopenic Purpura (ITP)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IgPro10_4001; 2011-000263-27 (EudraCT Number)
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Results first posted 2015-10-19 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2015-09

CONDITIONS: Immune Thrombocytopenic Purpura
Keywords: ITP
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IgPro10 (Experimental)
  Interventions: Biological: IgPro10

INTERVENTIONS:
Biological: IgPro10 — IgPro10 will be administrated by IV infusion either a single dose of 1 g/kg bw on 1 day or 2 doses of 1 g/kg bw on 2 days (2 g/kg bw total dose) dependent on the response to the first treatment.
  Other Names: Privigen

SUMMARY:
It is known that intravenous immunoglobulins can induce hemolysis, but the mechanism is not known in detail. The primary objective of this study was to investigate the specificity of antigens on red blood cells in patients with chronic immune thrombocytopenic purpura (ITP) who have shown signs of clinically relevant hemolysis following treatment with the intravenous immunoglobin Privigen®. The study was to explore potential mechanisms of hemolysis by analysis of the specificity of the antibodies possibly involved. To distinguish between clinically non-relevant hemolysis and a relevant intravascular hemolysis, an independent adjudication by a committee was performed for each patient with signs of hemolysis determined in the laboratory or in the clinic.

This study was requested as a post-marketing commitment study by the United States Food and Drug Administration (FDA). By September 2014, no case of clinically significant intravascular hemolysis was found, and the FDA agreed to halt the study and analyze all hemolysis-relevant endpoints using FDA criteria for hemolysis in addition to analyses planned in the protocol. The study was not restarted.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic ITP
* Age of 18 to 65 years
* Platelet count of ≤ 30 x 10^9/L at screening

Exclusion Criteria:

* Planned splenectomy throughout the study period
* Treatment with immunoglobulin G for intravenous administration (IVIG) or anti-D immunoglobulin within 3 weeks prior to screening
* Use of drugs that have any pharmacological effect on the blood clotting system within 3 weeks prior to screening
* Known allergy or other severe reactions to blood products including intolerability to previous IVIG
* Known hyperprolinemia
* Red blood cell transfusion or erythropoietin treatment within the last 14 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2011-11; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wieslaw Jedrzejczak, Principal Investigator — Samodzielny Publiczny Centralny Szpital Kliniczny w Warszawie
Locations (17):
- Bulgaria (3):
  - UMHAT "Dr. Georgi Stranski" Clinic of Haematology, Pleven
  - UMHAT "Sv. Georgi" Clinic of Haematology, Plovdiv
  - Tokuda Hospital, Sofia
- Romania (10):
  - Emergency Clinical County Hospital Baia Mare, Baia Mare
  - Emergency Clinical County Hospital Brasov, Brasov
  - Clinical Institute "Fundeni", Bucharest
  - Universitary Hospital, Bucharest
  - Clinical City Hospital "Filantropia", Craiova
  - City Hospital Oradea, Oradea
  - Emergency Clinical County Hospital Tg. Mures, Tg. Mures
  - Emergency Clinical City Hospital Timisoara, Timișoara
  - Oncomed SRL, Timișoara
  - Salvo-San-Ciobanca SRL, Zalău
- Serbia (4):
  - Clinical Center of Serbia, Belgrade
  - Clinical Hospital Bezanijska Kosa, Belgrade
  - Clinical Hospital Zemun, Belgrade
  - Clinical Center Nis, Niš

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Screening occurred within 6 days before treatment with IgPro10 (Privigen). Subjects who met all of the inclusion criteria and none of the exclusion criteria could be enrolled into the study. Of 58 eligible subjects, one withdrew consent before treatment and 57 subjects received at least 1 dose of Privigen.
Groups:
- IgPro10: IgPro10 was administered by IV infusion either as a single dose of 1 g/kg bw on 1 day or 2 doses of 1 g/kg bw on 2 days (2 g/kg bw total dose) dependent on the response to the first IgPro10 dose.
Period: Overall Study
Arm/Group | IgPro10
Started | 57 (Subjects treated with Privigen)
Completed | 56
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Subjects treated with Privigen
Arm/Group | IgPro10
Number analyzed (Participants) | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 55
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (13.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Set of Antibodies Most Frequently Bound to Red Blood Cells (RBCs) in Subjects Experiencing Clinically Significant Intravascular Hemolysis
Description: The occurrence of clinically significant intravascular hemolysis was determined by an independent Adjudication Committee. No subject experienced clinically significant intravascular hemolysis; therefore, the primary safety endpoint could not be analyzed.
Time Frame: Within 3 days of infusion
Arm/Group | IgPro10
Number analyzed (Participants) | 0

2. Secondary Outcome: Responder Rate
Description: The responder rate is the percentage of subjects who have a platelet response (defined as a platelet count increase at least once to ≥ 50 x 10^9/L after the first IgPro10 administration).
Time Frame: Within 6 days after the first infusion
Population: Full analysis set: all subjects who received at least 1 IgPro10 infusion.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IgPro10
Number analyzed (Participants) | 57
percentage of participants | 74 [61 to 83]

ADVERSE EVENTS:
Time Frame: For the duration of individual subject participation in the study, up to approximately 35 days.
Arm/Group | IgPro10
Serious Adverse Events (participants affected / at risk) | 1/57
Other Adverse Events (participants affected / at risk) | 19/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IgPro10 (N=57)
Immune Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IgPro10 (N=57)
Headache (Nervous system disorders) | 17 (23)
Pyrexia (General disorders) | 3 (6) — Adverse event collected under MedDRA 'General Disorders And Administration Site Conditions'.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CSL agreements and restrictions on publishing may vary with individual investigators; however, CSL will not prohibit any investigator from publishing. CSL supports the publication of results from all centers of a multi-center trial and generally requires that reports based on single-site data not precede the primary publication of the entire clinical trial.